CLINICAL TRIAL: NCT06822569
Title: Teen Health Choices & Wellness
Acronym: THC&W
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023003584; R01DA055600 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-02-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Health Behavior; Wellness, Psychological; Substance Use
MeSH Terms: conditions — Health Behavior; Psychological Well-Being; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Naturalistic, longitudinal (Other): Teenagers ages 13 to 16 years at the time of recruitment.
  Interventions: Other: Cue reactivity paradigm

INTERVENTIONS:
Other: Cue reactivity paradigm — Participants will be exposed to cues in a fixed sequence while they answer questions about their emotions and thoughts. The cues will include everyday items (e.g., an ink pen) and substance-related items (e.g., a vape pen).

SUMMARY:
The goal of this observational study is to learn more about changes in health, wellness, and substance-use behaviors as teenagers get older. Participants, ages 13 to 16, will be asked to use a smartphone application developed for this research study. Participants will also come to Brown University or meet via video conference to answer questions about specific behaviors, choices, and feelings that may change over time.

ELIGIBILITY:
Inclusion Criteria:

1. be age 13 to 16 years
2. engage in a target health behavior on at least one recent occasion
3. speak, read, and understand English or Spanish
4. live in or near Rhode Island

Exclusion Criteria:

1. lifetime history of moderate or severe substance use disorder or treatment, excluding nicotine use disorder
2. current psychotic symptoms or active suicidality (i.e., intent in the past 30 days)

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Maximum subjective craving during cannabis cue exposure (rated on a 0 to 10 scale). | Baseline, 1 year, 2 years
  This study utilizes a structured cannabis cue exposure paradigm. During cue exposure, participants rate subjective craving on a scale from 0, "Not at all," to 10, "Extremely." The specific item to assess positive effects is the question, "How strong is your craving to use cannabis right now" sourced from the Morean' Drug Craving Questionnaire-Now. See reference section.

SECONDARY OUTCOMES:
Maximum subjective positive effects of cannabis use in daily life (rated on a 0 to 10 scale). | Baseline, 1 year, 2 years
  This study utilizes a smartphone application to collect self-reported subjective cannabis effects in the participant's daily life. Following a self-initiated report of cannabis use in daily life, participants rate subjective positive effects of cannabis at that moment (i.e., "right now") on a scale from 0, "Not at all," to 10, "Extremely." The specific item to assess positive effects is the question, "Do you like any of the effects you are feeling right now?" sourced from the Tiffany's Drug Effects Questionnaire. See reference section.

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that cannot individually identify participants may be shared with researchers internal and external to Brown University upon reasonable request by qualified research collaborators. Data shared with qualified researchers will not contain any protected health information or other personally identifiable information that could be used to identify individual participants.

REFERENCES:
- [Background] Morean ME, de Wit H, King AC, Sofuoglu M, Rueger SY, O'Malley SS. The drug effects questionnaire: psychometric support across three drug types. Psychopharmacology (Berl). 2013 May;227(1):177-92. doi: 10.1007/s00213-012-2954-z. Epub 2012 Dec 28. PMID 23271193
- [Background] Tiffany ST, Singleton E, Haertzen CA, Henningfield JE. The development of a cocaine craving questionnaire. Drug Alcohol Depend. 1993 Dec;34(1):19-28. doi: 10.1016/0376-8716(93)90042-o. PMID 8174499